CLINICAL TRIAL: NCT03886259
Title: Effect of Neuromuscular Exercise in Combination With Pain Neuroscience Education Compared to Pain Neuroscience Education Alone in Patients With Chronic Pain After Primary Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Effects of Exercise and Education in Patients With Chronic Pain After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Northern Orthopaedic Division, Denmark (Other); The Danish Rheumatism Association (Other); Svend Andersen Foundation (Unknown); Lions Denmark (Unknown)
Responsible Party: Principal Investigator, Jesper Bie Larsen, PhD-student, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20180046
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Arthroplasty, Replacement, Knee; Chronic Pain
Keywords: Chronic Pain; Total Knee Arthroplasty; Pain Neuroscience Education; Neuromuscular exercise (NEMEX-TJR)
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded towards group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and pain neuroscience education (Experimental): Subjects with chronic pain after total knee replacement will receive 24 sessions of neuromuscular exercise therapy, supervised by a physiotherapist, and two sessions of pain neuroscience education, conducted by a physiotherapist
  Interventions: Other: Neuromuscular exercises (NEMEX-TJR) and pain neuroscience education
- Pain neuroscience education (Active Comparator): Subjects with chronic pain after total knee replacement will receive two sessions of pain neuroscience education, conducted by a physiotherapist
  Interventions: Other: Pain neuroscience education

INTERVENTIONS:
Other: Neuromuscular exercises (NEMEX-TJR) and pain neuroscience education — 60min. of neuromuscular exercises (NEMEX-TJR) training two times a week for 3 months (12 weeks, 24 sessions). Physiotherapists will instruct and supervise the participants during the neuromuscular exercises. The aim of the neuromuscular exercise program is to restore normal movement, improve sensorimotor control, re-establishing normal motor program strategies and muscle activation.
  60min. of pain neuroscience education at the beginning of intervention period and after 6 weeks. Both sessions will take 60min. and will be conducted by physiotherapists. The aim of the pain neuroscience education is to increase the pain neuroscience knowledge of the patients leading to a better understanding of their chronic pain and thereby engaging the patients in the treatment of their chronic pain and impaired function.
  Arms: Exercise and pain neuroscience education
Other: Pain neuroscience education — 60min. of pain neuroscience education at the beginning of intervention period and after 6 weeks. Both sessions will take 60min. and will be conducted by physiotherapists. The aim of the pain neuroscience education is to increase the pain neuroscience knowledge of the patients leading to a better understanding of their chronic pain and thereby engaging the patients in the treatment of their chronic pain and impaired function.
  Arms: Pain neuroscience education

SUMMARY:
The purpose of the study is to investigate whether a 12-week neuromuscular rehabilitation program (NEMEX-TJR) combined with pain neuroscience education (PNE) provides greater pain relief, improvement in physical function and quality of life than PNE alone in a population of patients with chronic pain after primary total knee arthroplasty.

Hypothesis: Rehabilitation involving neuromuscular training and PNE will provide greater pain relief, improved function and improved quality of life compared to PNE alone at the primary endpoint, which is follow-up 12months after the start of the treatment.

DETAILED DESCRIPTION:
Osteoarthritis is considered the most frequent cause of disability and pain in the elderly population, and the knee joint is one of the joints most commonly affected.

End-stage osteoarthritis is often treated with knee replacement, and total knee arthroplasty is considered an effective treatment for pain relief and improved function. However, several studies have reported less favorable outcomes after total knee arthroplasty, and systematic reviews found chronic pain after total knee arthroplasty at 12 months post-operative in 13-17% of the patients and chronic pain rates at 2-7 years post-operative varying between 8-27%. No randomized controlled trials evaluating exercise and pain education treatments to patients with chronic pain after total knee arthroplasty exists, and this highlights the need for evidence-based knowledge of which treatment should be considered for this population.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 19-40
* Subjects with primary total knee arthroplasty due to osteoarthritis ≥ 12 months post-operatively
* For the index knee, duration of knee pain > 6 months
* For the index knee, the average daily pain score ≥ 4 (moderate-to-severe pain) over the last week prior to visit on a numeric rating scale

Exclusion Criteria:

* Specific reasons for chronic pain, such as loosening of implant, which requires revision surgery
* Secondary causes of arthritis to the knee, e.g. rheumatoid arthritis
* Surgery (including arthroscopy) of the index knee within 3 months prior to visit
* Injury to the index knee within 12 months prior to visit
* Recent history of acute pain affecting the lower limb and/or trunk
* Participation in other pain trials two weeks prior to this study
* Pregnancy
* Drug and alcohol abuse
* Previous neurologic illnesses or primary pain area other than knee, e.g. lower back, upper extremity pain or rheumatoid arthritis
* Lack of ability to adhere to protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score4 (KOOS4) from baseline to 12months follow-up | Baseline and at 3, 6 and 12 months
  The average score for four of the five KOOS subscales, covering pain, symptoms, difficulties in functions of daily living, and quality of life (KOOS4), with scores ranging from 0 (worst) to 100 (best). Between group comparisons of treatment effect (change in KOOS4 from baseline to 1 year follow-up) will be performed.

SECONDARY OUTCOMES:
Change in all five subscales of the KOOS | Baseline and at 3, 6 and 12 months
  All five domains, covering pain, symptoms, difficulties in functions of daily living, sport and recreation and quality of life of the questionnaire will be used as secondary outcome with scores ranging from 0 (worst) to 100 (best).
Rating of Global Perceived Effect | 3, 6 and 12 months
  Global Perceived Effect will be assessed using the question: "How are your knee problems now compared with before you entered this study"? The question will be answered on a seven-point Likert scale ranging from 'Improved, an important improvement' to 'Worse, an important worsening'.
Change in maximal pain intensity during rest (day and night), stair climbing, and walking on a Numeric Rating Scale (NRS) | Baseline and at 3, 6 and 12 months
  Pain intensities on a NRS, where "0" represents "no pain" and "10" represents "maximal pain" in various situations.
Change in use of Pain Medication | Baseline and at 3, 6 and 12 months
  Dosage of pain medication used within last week
Number of adverse events related to interventions | 3 months
  Serious and non-serious events that may occur during the intervention period will be identified in different ways: by self-reporting by the participants and by observation from the physiotherapists. Adverse events will be categorized as occurring in the index knee or other sites than the index knee.
Change in 40-meter fast-paced walk test | Baseline and at 3, 6 and 12 months
  The amount of time in seconds it takes to complete the 40m
Change in stair climb test | Baseline and at 3, 6 and 12 months
  The amount of time in seconds it takes to complete ascending and descending of 9 stairs
Change in 30-second chair stand test | Baseline and at 3, 6 and 12 months
  Number of repetitions in 30-seconds
Change in PainDETECT scores | Baseline and at 3, 6 and 12 months
  The questionnaire is comprised of 3 major components: graduation of pain, pain course pattern and radiating pain. The maximum possible score is 38, and the minimum possible score is -1.
Change in score from the Fear-avoidance Beliefs Questionnaire - Physical Activity | Baseline and at 3, 6 and 12 months
  The scores range from "0" with "completely disagree" to "6" with "completely agree" and sums up to a total score between 0-24.
Change in score from the Pain Catastrophizing Scale | Baseline and at 3, 6 and 12 months
  Scores is rated on a 5-point scale with the 0 being "not at all" and 4 being "all the time" and the score can range from 0 to 52 points.
Change in pinprick hyperalgesia at index knee and extrasegmental | Baseline and at 3, 6 and 12 months
  The subject is to rate the pain intensity from the pinprick on a NRS, where "0" represents "no pain" and "10" represents "maximal pain".
Change in temporal summation at index knee and extrasegmental | Baseline and at 3, 6 and 12 months
  The subject is to rate the pain intensity of the last test stimulus on a NRS, where "0" represents "no pain" and "10" represents "maximal pain".
Change in dynamic mechanical allodynia at the index knee and extrasegmental | Baseline and at 3, 6 and 12 months
  The subject is to rate the pain intensity of a cotton swab on a NRS, where "0" represents "no pain" and "10" represents "maximal pain".
Change in deep somatic hyperalgesia at the index knee and extrasegmental | Baseline and at 3, 6 and 12 months
  A "bedside algometer" will be applied on the skin over the vastus medialis muscle on the index side. The subject is to indicate immediately when the pressure becomes painful.
Change in pressure pain thresholds at the index knee and extrasegmental | Baseline and at 3, 6 and 12 months
  Pressure pain thresholds measured using a handheld algometer (Algometer Type II, Somedic AB, Hoerby, Sweden)) at the index knee and extrasegmental.
Change in descending pain control | Baseline and at 3, 6 and 12 months
  Conditioned pain modulation effect will be measured comparing the test stimuli without conditioning stimuli to the test stimuli with conditioning stimuli
Change in number of sites with usual pain shaded on a body chart | Baseline and at 3, 6 and 12 months
  Shaded markings on a body chart to indicate where usual pain is located
Change in leg extension power | Baseline and at 3, 6 and 12 months
  Leg extension power in a single-leg simultaneous hip and knee extension will be measured bilaterally. Highest measurement in watt is the outcome.
Change in isometric muscle strength of knee extensors and flexors | Baseline and at 3, 6 and 12 months
  Maximum isometric muscle strength (measured in Newtons) measured bilaterally in knee flexion and knee extension in a test using a handheld dynamometer (Lafayette manual muscle tester from Lafayette Instruments, USA).

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale | Baseline
  The questionnaire consists of 14 items, which measures the patient level of anxiety and depression. The score in each item ranges from 0-3, giving scoring ranges from 0-21.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Madeleine, Dr.Scient, Study Chair — Aalborg University; Søren T Skou, PhD, Study Chair — University of Southern Denmark and Næstved-Slagelse-Ringsted Hospitals; Ole Simonsen, Dr.Med, Study Chair — Aalborg University Hospital; Lars Arendt-Nielsen, Dr.Med, Study Chair — Aalborg University; Jesper B Larsen, M.Sc., Principal Investigator — Aalborg University; Mogens B Laursen, PhD, Study Chair — Aalborg University Hospital
Locations (3):
- Denmark (3):
  - Department of Occupational and Physiotherapy, Aalborg University Hospital, Aalborg
  - Department of Occupational- and Physiotherapy, Aalborg University Hospital, Farsø
  - Department of Occupational- and Physiotherapy, Aalborg University Hospital, Thisted

IPD SHARING:
Plan to Share IPD: Yes
Individual subject data that underlie the results reported in the publication will be shared after deidentification (text, tables, figures, appendices)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months following publication. No end date.
Access Criteria: Researchers that provide a methodologically sound plan

REFERENCES:
- [Background] Peat G, McCarney R, Croft P. Knee pain and osteoarthritis in older adults: a review of community burden and current use of primary health care. Ann Rheum Dis. 2001 Feb;60(2):91-7. doi: 10.1136/ard.60.2.91. PMID 11156538
- [Background] Dieppe PA, Lohmander LS. Pathogenesis and management of pain in osteoarthritis. Lancet. 2005 Mar 12-18;365(9463):965-73. doi: 10.1016/S0140-6736(05)71086-2. PMID 15766999
- [Background] Davidson D, de Steiger R, Graves S, Tomkins A et al. Australian orthopaedic association national joint replacement registry. annual report. Adelaide:AOA;2010. . 2010
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Bhave A, Mont M, Tennis S, Nickey M, Starr R, Etienne G. Functional problems and treatment solutions after total hip and knee joint arthroplasty. J Bone Joint Surg Am. 2005;87 Suppl 2:9-21. doi: 10.2106/JBJS.E.00628. No abstract available. PMID 16326719
- [Background] Wylde V, Dieppe P, Hewlett S, Learmonth ID. Total knee replacement: is it really an effective procedure for all? Knee. 2007 Dec;14(6):417-23. doi: 10.1016/j.knee.2007.06.001. Epub 2007 Jun 26. PMID 17596949
- [Background] Beswick AD, Wylde V, Gooberman-Hill R, Blom A, Dieppe P. What proportion of patients report long-term pain after total hip or knee replacement for osteoarthritis? A systematic review of prospective studies in unselected patients. BMJ Open. 2012 Feb 22;2(1):e000435. doi: 10.1136/bmjopen-2011-000435. Print 2012. PMID 22357571
- [Background] Wylde V, Dennis J, Beswick AD, Bruce J, Eccleston C, Howells N, Peters TJ, Gooberman-Hill R. Systematic review of management of chronic pain after surgery. Br J Surg. 2017 Sep;104(10):1293-1306. doi: 10.1002/bjs.10601. Epub 2017 Jul 6. PMID 28681962
- [Background] Beswick AD, Wylde V, Gooberman-Hill R. Interventions for the prediction and management of chronic postsurgical pain after total knee replacement: systematic review of randomised controlled trials. BMJ Open. 2015 May 12;5(5):e007387. doi: 10.1136/bmjopen-2014-007387. PMID 25967998
- [Background] Larsen JB, Skou ST, Arendt-Nielsen L, Simonsen O, Madeleine P. Neuromuscular exercise and pain neuroscience education compared with pain neuroscience education alone in patients with chronic pain after primary total knee arthroplasty: study protocol for the NEPNEP randomized controlled trial. Trials. 2020 Feb 24;21(1):218. doi: 10.1186/s13063-020-4126-5. PMID 32197629
- [Derived] Larsen JB, Skou ST, Laursen M, Bruun NH, Arendt-Nielsen L, Madeleine P. Exercise and Pain Neuroscience Education for Patients With Chronic Pain After Total Knee Arthroplasty: A Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e2412179. doi: 10.1001/jamanetworkopen.2024.12179. PMID 38787559

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT03886259/SAP_000.pdf